CLINICAL TRIAL: NCT01284153
Title: A Comparison of Three Radiotherapy Techniques for Breast Cancer: a Planning Study
Brief Title: Potential Benefits of Radiotherapy in Prone Position for Breast Cancer Patients: a Planning Study
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof. Caroline Weltens, UZ Leuven
Other Study IDs: S52869
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms; Radiation
Keywords: respiratory gating; prone radiotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study has the purpose to investigate the benefit of treating breast cancer patients in prone position. This treatment is compared to the standard technique in our center (supine position with or without respiratory gating). The investigators want to compare the doses on the organs at risk (heart and lungs) in the different techniques.

ELIGIBILITY:
Inclusion Criteria:

* indication for radiotherapy of the breast and /or lymph nodes

Exclusion Criteria:

* none ( planning study)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have an indication for radiotherapy of the breast and/or the lymph nodes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Sweldens, Doctor, Study Director — UZ Leuven
Locations (1):
- UZ Leuven Radiotherapy Department, Leuven, Belgium